CLINICAL TRIAL: NCT00707837
Title: Effect of Supplemental Infant Formula on Blood Levels in Preterm Infants
Brief Title: Nutritional Study in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK15
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2008-09

CONDITIONS: Preterm Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infant Formula (Experimental): Preterm infant formulas containing lipid soluble compounds
  Interventions: Other: Preterm infant formula with added soluble lipids
- Preterm formulas (Active Comparator): Standard preterm infant formula and discharge formulas
  Interventions: Other: Preterm infant formulas and discharge formulas

INTERVENTIONS:
Other: Preterm infant formulas and discharge formulas — Preterm infant formulas to be consumed per health care provider orders
  Arms: Preterm formulas
Other: Preterm infant formula with added soluble lipids — Preterm infant formula to be fed per healthcare provider instructions
  Arms: Infant Formula

SUMMARY:
An evaluation of a preterm infant formula containing ingredients similar to those found in breastmilk

ELIGIBILITY:
Inclusion Criteria:

* Birthweight 500-1800 g
* Less than 33 wks gestational age
* Enteral feeding initiated by 21 days of life
* Asymmetrical small-for-gestational age (SGA) infants and infants with patent ductus arteriosus (PDA) are eligible to participate
* Singleton or twin births only
* Infant is 21 days of age or less at time of randomization

Exclusion Criteria:

* Serious congenital abnormalities that may affect growth and development
* Grade III or IV intraventricular hemorrhage (IVH)
* Maternal incapacity
* History of major surgery
* Extracorporeal membrane oxygenation (ECMO)
* Asphyxia
* Confirmed NEC or positive blood cultures at the time of randomization

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the serum concentrations of fat soluble compounds in preterm infants fed a regimen of preterm formulas and in human milk fed infants | variable

SECONDARY OUTCOMES:
Measures of eye function, ROP, measures of skin lipid soluble compound concentration | variable

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Barrett-Reis, PhD, Study Chair — Abbott Nutrition
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - West Coast Neonatalogy, All Children's Hospital, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - Maria Fareri Children's Hospital at Winchester Medical Center, Vahalla, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah